CLINICAL TRIAL: NCT02628353
Title: Randomized, Cross-over, Double Blinded, Placebo-controlled Study for the Evaluation of the Postprandial Effect of a Specific PHENOLic Compound on Blood PRESSure
Brief Title: Effect of a Specific Phenolic Compound on Blood Pressure
Acronym: PHENOLPRESS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: University Rovira i Virgili (Other); Hospital Universitari Sant Joan de Reus (Other); Fundació Catalana per a la Recerca i la Innovació (FCRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LLAVOR 2014-00081
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Risk Factors; Blood Pressure
Keywords: Cardiovascular diseases; endothelial function; systolic blood pressure; metabolomics; cardiovascular risk factor; bioavailability; phenolic compounds; hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): control group
  Interventions: Dietary Supplement: placebo
- Phenolic compound (Experimental): treated group
  Interventions: Dietary Supplement: phenolic compound

INTERVENTIONS:
Dietary Supplement: placebo — 1 capsule of placebo product (100 mg carboxymetylcellulose) in one visit
  Arms: Placebo
Dietary Supplement: phenolic compound — 1 capsule of phenolic compound product (100mg phenolic compound + 100 mg carboxymetylcellulose) in one visit
  Arms: Phenolic compound

SUMMARY:
The study's main objective is to investigate the effects of acute consumption of a preparation containing 100 mg of a specific phenolic compound (patent pending, P201531587) on systolic BP after ingestion of a high fat meal.

DETAILED DESCRIPTION:
The study's main objective is to investigate the effects of acute consumption of a preparation containing 100 mg of a specific phenolic compound (patent pending, P201531587) on systolic blood pressure (BP) after ingestion of a high fat meal.

The secondaries objectives are:

* To evaluate the effects on diastolic BP.
* To study the phenolic compound bioavailability and to analyze its metabolites for determine the phenolic compound consumption biomarkers.
* To evaluate the effects on endothelial function by ischemic reactive hyperemia (IRH).

The sample size was calculated using a previous studies using systolic blood pressure (SBP) as the primary outcome measure. A total of 14 subjects are needed, assuming variance components of approximately 20.0, to detect differences between treatments (placebo and phenolic product) of 10 mmHg, with a bilateral significance level of α=0.05, a power of 80% and a standard deviation of 11.82 mmHg at the baseline.

To compare the main variable efficiency of the products of study as well as secondary variables of efficiency, will carry out analysis of the covariance (ANCOVA) with basal value as covariable, followed by the Tukey test for determining multiple differences. All tests will be carried out with significance to bilateral level of 5%. It is considered significant value p<0,05. The data will be analyzed using the "SPSS" program version 22.

The statistical analysis will follow the principles specified in the guidelines of the International Conference on Harmonization (ICH) E9 and CPMP/EWP/908/99 ICH E9 Points to Consider on Multiplicity Issues in Clinical Trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults men or women (>18 years old)
* Blood pressure (with no drug intervention) ≥130 mm Hg systolic blood pressure ≤ 159 mmHg
* No evidence of chronic disease
* Written informed consent provided before the initial screening visit.

Exclusion Criteria:

* Systolic blood pressure ≥ 160 mm Hg and diastolic blood pressure ≥100 mm Hg or taking antihypertensive medication
* Body mass index (BMI) ≥ 35 kg/m2
* Glucose (fasting state) >125 mg/dL
* LDL-cholesterol >189 mg/dL
* Triglycerides >350 mg/dL
* Pregnant or intending to become pregnant
* Use of medication, antioxidant, or multi-vitamin supplements
* Chronic alcoholism
* Intense physical activity (5h/week)
* Intestinal disorders
* Following of a vegetarian diet
* Anemia (hemoglobin ≤13 g/dL in men and ≤12 g/dL in women)
* Being intolerant or suffer from allergy to any of the products of the high fat meal (white bread, olive oil, boiled egg, cheese) or to the products of the study.
* Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study.
* Failure to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change of Systolic Blood Pressure | In each visit (2 visits in total), systolic blood pressure will be measured at baseline (0 min) and 60, 120, 180, 240, 300 and 360 minutes after the ingestion of a fat load and the supplement.
  During each visit (2 visits in total), systolic BP will be measured after 10 min in a seated position in a comfortable room by the physician. The measurement will be taken in triplicate at 1-min intervals using an automatic sphygmomanometer (OMRON HEM-907; PEROXFARMA, Barcelona, Spain). The first measurement will be discarded and the final result will be the average of the other measurements..
  The research team will mesure the change in the evolution of systolic blood pressure between visits (at least 1 week between visits).

SECONDARY OUTCOMES:
Diastolic Blood Pressure | In each visit (2 visits in total), diastolic blood pressure will be measured at baseline (0 min) and 60, 120, 180, 240, 300 and 360 minutes after the ingestion of a fat load and the supplement.
  During each visit (2 visits in total), diastolic BP will be measured after 10 min in a seated position in a comfortable room by the physician. The measurement will be taken in triplicate at 1-min intervals using an automatic sphygmomanometer (OMRON HEM-907; PEROXFARMA, Barcelona, Spain). The first measurement will be discarded and the final result will be the average of the other measurements..
  The research team will mesure the change in the evolution of diastolic blood pressure between visits (at least 1 week between visits).
Ischemic reactive hyperemia (IRH) | In each visit (2 visits in total), at 0, 120, 240 and 360 minutes
  The endothelial-dependent vasomotor functions will be measured as IRH by a Laser-Doppler linear PERIFLUX 5000 flowmeter (PERIMED AB, Stockholm, Sweden)
Bioavailability of phenolic compound in plasma samples | In each visit (2 visits in total), at 0, 60, 120, 180, 240, 300 and 360 minutes (heparin lithium plasma)
  The phenolic compound bioavailability will be analysed in all volunteers and according to the technical reference at the time of its determination, as it may be to analyse automatic, ELISA kits, or other techniques.
Bioavailability of phenolic compound in urine | In each visit (2 visits in total), at 0, 180 and 360 minutes (total urine)
  The phenolic compound bioavailability will be analysed according to the technical reference at the time of its determination, as it may be to analyse automatic, ELISA kits, or other techniques

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, PhD, Principal Investigator — University Rovira i Virgili / Hospital Universitari Sant Joan de Reus; Begoña Muguerza, PhD, Study Chair — University Rovira i Virgili
Locations (1):
- Technological Centre of Nutrition and Health (CTNS), Reus, Tarragona, Spain

REFERENCES:
- See also: Technological Centre of Nutrition and Health — http://www.ctns.cat/en